CLINICAL TRIAL: NCT01665261
Title: Accuracy Assessment of 7 Clinical Indicators in Newborn Screening for Congenital Heart Disease
Brief Title: Newborn Screening for Congenital Heart Disease
Acronym: NSCHD
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Guoying huang, President of Children's Hospital of Fudan University, Fudan University
Other Study IDs: KY2011-366-1
Record Dates: First submitted 2012-08-09; First posted 2012-08-15 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; Newborn; Pulse oximetry; Screening
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to test the accuracy of 7 indicators in screening congenital heart defects (CHD) in all newborns (symptomatic or asymptomatic) to determine whether these indicators could be applied in the nationwide newborn CHD screening. The investigator's hypothesis is that 7 indicators are effective in neonate CHD screening with the acceptable accuracy.

DETAILED DESCRIPTION:
Congenital heart defects (CHD) are among the most common major congenital anomalies, and they occur worldwide with an incidence of about 8-12/1,000 live births , Most of these defects are mild or moderate. They either do not need treatment or treatment is needed only after infancy. Other defects are severe and require early treatment in infancy, which are the primary objectives of screening, because they are at risk of adverse or irreversible outcomes as a consequence of congenital heart defects. However, about half the neonates in the nursery have no distinctive clinical signs (symptoms, abnormal murmurs or cyanosis).So it's necessary to develop a screening strategy for neonatologist and pediatrician, especially physicians in community. Screening strategy in our study consists of 7 indicators: Family history of CHD, tachypnea, heart murmurs(≥ 2 grade), cyanosis, other non-cardiac malformations,special face feature（relating to chromosomal or non-chromosomal syndromes）, subnormal Pulse Oximetry reading (Oxygen saturation of less than 95% in either limb or more than 3% difference）。The newborn babies with any of these 7 indicators positive will be considered positive-screened and echocardiography will performed.

The whole study (screening for CHDs with 7 indicators and performing the echocardiography for diagnosis) will be conducted by one single investigator (Quming Zhao from Children's Hospital of Fudan University). The new generation Pulse Oximetry has been proved to have low intraobserver and interobserver variability, but the interobserver variability in clinical evaluation (especially murmurs and cyanosis) remain unknown, the investigator will also assess the interobserver variability by comparing Quming Zhao and other two pediatricians (from the participating Hospital)(blind to each other).

ELIGIBILITY:
Inclusion Criteria:

* all consecutive live newborn infants
* between 6-72hours of age

Exclusion Criteria:

* declining the screening;
* early discharge before the screening;
* missing

Ages: 6 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All consecutive neonates including pre-mature neonates and symptomatic neonates) will be recruited prospectively from two collaboration hospitals of the ongoing projects- "Key Clinical Research Project Sponsored by Ministry of Health Screening, evaluation and intervention of congenital heart disease in newborn infants(2010-239)"
Sampling Method: Probability Sample
Enrollment: 6730 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the 7 indicators for detection of all CHDs and major CHDs | The goldstandard for CHD diagnosis is the echocardiography performed within 1 hour from the screening completed.
  Sensitivity, specificity, negative and positive predictive value, negative and positive likelihood ratio of 7 indicators for the detection of all CHDs and major CHDs as gold standard the echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Huang G Ying, MD PHD, Study Chair — Children's Hospital of Fudan University
Locations (2):
- China (2):
  - Songjiang District Central Hospital, Shanghai, Shanghai Municipality
  - Songjiang Maternal and Child Health Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] de-Wahl Granelli A, Wennergren M, Sandberg K, Mellander M, Bejlum C, Inganas L, Eriksson M, Segerdahl N, Agren A, Ekman-Joelsson BM, Sunnegardh J, Verdicchio M, Ostman-Smith I. Impact of pulse oximetry screening on the detection of duct dependent congenital heart disease: a Swedish prospective screening study in 39,821 newborns. BMJ. 2009 Jan 8;338:a3037. doi: 10.1136/bmj.a3037. PMID 19131383
- [Background] Ewer AK, Furmston AT, Middleton LJ, Deeks JJ, Daniels JP, Pattison HM, Powell R, Roberts TE, Barton P, Auguste P, Bhoyar A, Thangaratinam S, Tonks AM, Satodia P, Deshpande S, Kumararatne B, Sivakumar S, Mupanemunda R, Khan KS. Pulse oximetry as a screening test for congenital heart defects in newborn infants: a test accuracy study with evaluation of acceptability and cost-effectiveness. Health Technol Assess. 2012;16(2):v-xiii, 1-184. doi: 10.3310/hta16020. PMID 22284744
- [Background] Mahle WT, Newburger JW, Matherne GP, Smith FC, Hoke TR, Koppel R, Gidding SS, Beekman RH 3rd, Grosse SD; American Heart Association Congenital Heart Defects Committee of the Council on Cardiovascular Disease in the Young, Council on Cardiovascular Nursing, and Interdisciplinary Council on Quality of Care and Outcomes Research; American Academy of Pediatrics Section on Cardiology and Cardiac Surgery, and Committee on Fetus and Newborn. Role of pulse oximetry in examining newborns for congenital heart disease: a scientific statement from the American Heart Association and American Academy of Pediatrics. Circulation. 2009 Aug 4;120(5):447-58. doi: 10.1161/CIRCULATIONAHA.109.192576. Epub 2009 Jul 6. PMID 19581492